CLINICAL TRIAL: NCT04421014
Title: Ketone Ester Effects on Biomarkers of Brain Metabolism and Cognitive Performance in Cognitively Intact Adults >= 55 Years Old. A Double-Blinded Randomized Controlled Clinical Trial.
Brief Title: Ketone Ester Effects on Biomarkers of Brain Metabolism and Cognitive Performance in Cognitively Intact Adults 55 Years Old or Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200087; 20-AG-0087
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06-02

CONDITIONS: Metabolic Syndrome; Normal Cognition
Keywords: Ketogenic; Brain Metabolism; BETA-HYDROXYBUTYRATE; Dietary Supplement; Alzheimer's Disease
MeSH Terms: conditions — Metabolic Syndrome; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone Ester drink/ Arm 1 (Active Comparator): 25 participants
  Interventions: Dietary Supplement: Ketone Ester drink
- Placebo/ Arm 2 (Placebo Comparator): 25 participants
  Interventions: Dietary Supplement: Placebo: isocaloric dextrose drink

INTERVENTIONS:
Dietary Supplement: Ketone Ester drink — The main ingredient of the Ketone Ester drink [(R)-3-hydroxybutyl (R)-3-hydroxybutyrate)] is regulated as GRAS (Generally Recognized as Safe) substance by the FDA (https://www.accessdata.fda.gov/scripts/fdcc/index.cfm?set=GRASNotices&id=515). The Ketone Ester compound is already being sold in the market as a ketogenic supplement and is especially popular among athletes, such as cyclists (sold by the official website of the company TdeltaS(R) Global (https://www.deltagketones.com/products/g-ketone-performance). The dose and formulation (25 g of KE contained in 59 ml of a drink), daily scheme (3 times daily) and total duration (28 days) are identical to a previous safety human study. The Ketone Ester drink provided by DeltaG will be repackaged by the NIA Pharmacist into new bottles identical to the ones that will be used for the placebo to ensure the blinding of participants and researchers to the drink.
  Arms: Ketone Ester drink/ Arm 1
Dietary Supplement: Placebo: isocaloric dextrose drink — The main content of the Placebo will be an aqueous solution containing approximately 35 g of dextrose, a fruity flavor powder and stevia. We will also add Denatonium Benzoate (Bittrex) to match the bitterness of the Ketone Ester drink. The placebo will be prepared and dispensed by the NIA Pharmacist.
  Arms: Placebo/ Arm 2

SUMMARY:
Background:

In Alzheimer s disease (AD) the brain cannot use glucose as a fuel. The brain can use ketones as a fuel instead of glucose. Researchers want to test a supplement, Ketone Ester (KE). It may improve brain metabolic function and cognition in normal people and, perhaps, down the road, in patients with AD.

Objective:

To study the change in brain ketone levels in people after 28 days of taking KE compared with baseline and placebo. Also, to study changes in cognitive performance.

Eligibility:

People 55 years old or older with metabolic syndrome and no cognitive impairment

Design:

Participants will have 4 visits.

Participants will be screened at Visit 1 with:

Medical history

Physical exam

Blood and urine tests

Cognitive testing

Participants will be randomly assigned to receive either the study supplement or a placebo with same amount of calories. Neither they nor the researchers will know which they receive.

Visit 2 will include repeats of some screening tests. It will also include:

Stool sample (brought from home)

MRI/MRS: Participants will lie on a table that slides in and out of a scanner. A coil will be placed over their head. They may be asked to perform leg exercises.

First dose of study supplement or placebo

About 2 weeks after Visit 2, Visit 3 will include blood and urine tests and a questionnaire.

About 2 weeks after Visit 3, Visit 4 will include repeats of the Visit 2 tests.

Participants will drink the study supplement or placebo 3 times per day during the study. They will keep a daily log of each dose. They will bring the log to Visits 3 and 4.

Participants will by contacted by phone once per week during the study to see how they are doing.

...

DETAILED DESCRIPTION:
Study Description:

We hypothesize that supplementation with a ketone ester drink [Ketone Ester (KE)] compared to placebo, in cognitively intact adults >= 55 years old with Metabolic Syndrome (MetS), will (i) increase peripheral and brain ketone levels [primarily beta-hydroxybutyrate (BHB) and secondarily acetoacetate (AcAc)], (ii) improve neuronal/astrocytic insulin resistance (IR) and induce a change in neuronal/astrocytic metabolism as reflected on blood Extracellular Vesicle (EV) biomarkers, (iii) improve cognitive performance, (iv) boost mitochondrial function in muscle, and (v) change gut microbiome. These effects will be examined acutely, after single-dose administration, and chronically, after 28 days on the supplement x 3 times per day. The changes in EV biomarkers and cognition will be associated with the elevation of ketones in brain. The study will involve a Screening Visit and three additional Visits to assess acute effects, compliance and chronic effects, respectively, and a follow-up visit to obtain DNA.

Objectives:

Primary: To investigate the change in brain concentration BHB, using brain Magnetic Resonance Spectroscopy, after 28 days of supplementation with the KE, compared to baseline and placebo.

Secondary: To test the hypothesis that genetic factors may affect the response to the KE supplement.

Endpoints: Primary: To detect with brain MRS, a significant change in the concentration of BHB, after 28 days of supplementation with the KE compared to baseline and placebo

Secondary: To assess whether genetic factors modulate the response to the KE supplement.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to provide informed consent and willingness to sign a written informed consent document
2. Male or female, age >=55 years old
3. Cognitively intact status ascertained during screening (defined as absence of significant memory or cognitive changes in the last 2 years by subjective report, Clinical Dementia Rating (CDR) of 0, and Montreal Cognitive Assessment (MoCA) >= 26)
4. Ability to take oral medications
5. Willingness to adhere to all study procedures including having MRI/MRS.
6. Presence of Metabolic Syndrome (MetS). Specifically, they should meet three of the five following MetS diagnostic criteria to be eligible:

   * Receive drug treatment for elevated triglycerides (TGs) or have serum TGs >=150 mg/dL (1.7 mmol/L)
   * Receive drug treatment for low HDL-cholesterol or have serum HDL-cholesterol <40 mg/dL (1.0 mmol/L) in males; <50 mg/dL (1.3 mmol/L) in females
   * Receive drug treatment for high Blood Pressure (BP) or have BP >=130/85 mmHg
   * Receive drug treatment for high blood glucose or have fasting plasma glucose >=100 mg/dL
   * Central obesity, defined as a waist circumference >=102 cm (40 in) in men and >=88 cm (35 in) in women.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Previously diagnosed with a condition causing clinically significant cognitive impairment, such as MCI, AD or other type of dementia (such as vascular dementia, Lewy body dementia and frontotemporal dementia).
2. History of clinically significant brain disorders, such as stroke, multiple sclerosis, Parkinson s disease or other movement disorders, brain tumors, history of meningitis or encephalitis, history of moderate or severe traumatic brain injury (defined as Glasgow Coma Scale of 12 or less), epilepsy. Certain common neurological disorders not considered relevant (e.g. migraine, essential tremor) or incidental neuroimaging findings that are common and of uncertain clinical significance (e.g. mild-moderate microvascular changes on MRI) may be allowed.
3. Chronic and significant psychiatric conditions (e.g. history of bipolar disorder, schizophrenia, PTSD, moderate to severe depression or treatment-resistant depression. Unipolar depression or anxiety disorder may be allowed if mild or if successfully treated with single anti-depressant or anti-anxiety agents.
4. Positive urine drug screen (and no prescription medication accounting for the positive test).
5. Positive HIV, HBV or HCV status during screening.
6. Contraindications for MRI (pregnancy, pacemakers or other implanted devices, ferrous metal implants or shrapnel in or around the head etc.).
7. Anemia (defined as HGB < 12 for men or < 11 g/dl for women)
8. Poor venous access.
9. Lactation or Pregnancy (positive urine pregnancy test. Pregnancy tests will not be done on post-menopausal women defined as one of the below criteria:

   1. prior bilateral oophorectomy
   2. Amenorrhea for 12 months or more
10. Known severe allergic reactions to the KE drinks or other ketogenic supplement or stevia products.
11. Following high fat/low carb diet (ketogenic) diet or very low calorie (<500 calories) diet or taking other ketogenic supplements (such as Medium Chain Triglycerides (MCTs), Ketone Salts) or fasting intermittently and unwilling to stop it while on the KE drink/Placebo.
12. Very high or severe hypertriglyceridemia (>=886 mg/dL or 10.0 mmol/L)
13. Severe Hypertension (systolic blood pressure >=180 mmHg and/or diastolic blood pressure >=120 mmHg)
14. Weight >= 300 lbs (MRI scanner weight limit)
15. Diabetes Mellitus (type 1 or 2)
16. Taking the drug metformin.
17. Non-English speakers (given staffing constraints for cognitive testing administration and need for decreased variability in testing procedures for a small N study).
18. Participant has any concurrent medical condition, so that participation in the clinical study would not be in her/his best interest, in the PI s judgement.
19. To be eligible to consent for optional thigh MRI: Individuals with joint replacements that may be affected by the defined exercise protocol or which may prevent MRI analysis or any condition, in the opinion of the investigator, that would prevent successful completion of the exercise protocol such as, but not limited to reported osteoarthritis, rheumatoid arthritis and/or fibromyalgia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Brain concentration of BHB using brain Magnetic Resonance Spectroscopy | 28 days - outcome assessed at Visit 2 (baseline measurement before the first dose and after 75 min); Visit 4 (before and after 75 min from last dose).
  To detect with brain MRS, a significant change in the concentration of BHB, after 28 days of supplementation with the Ketone Ester drink compared to baseline and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios I Kapogiannis, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- [Background] Fortier M, Castellano CA, Croteau E, Langlois F, Bocti C, St-Pierre V, Vandenberghe C, Bernier M, Roy M, Descoteaux M, Whittingstall K, Lepage M, Turcotte EE, Fulop T, Cunnane SC. A ketogenic drink improves brain energy and some measures of cognition in mild cognitive impairment. Alzheimers Dement. 2019 May;15(5):625-634. doi: 10.1016/j.jalz.2018.12.017. Epub 2019 Apr 23. PMID 31027873
- [Background] Soto-Mota A, Vansant H, Evans RD, Clarke K. Safety and tolerability of sustained exogenous ketosis using ketone monoester drinks for 28 days in healthy adults. Regul Toxicol Pharmacol. 2019 Dec;109:104506. doi: 10.1016/j.yrtph.2019.104506. Epub 2019 Oct 23. PMID 31655093
- [Background] Cunnane SC, Courchesne-Loyer A, Vandenberghe C, St-Pierre V, Fortier M, Hennebelle M, Croteau E, Bocti C, Fulop T, Castellano CA. Can Ketones Help Rescue Brain Fuel Supply in Later Life? Implications for Cognitive Health during Aging and the Treatment of Alzheimer's Disease. Front Mol Neurosci. 2016 Jul 8;9:53. doi: 10.3389/fnmol.2016.00053. eCollection 2016. PMID 27458340
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-AG-0087.html